CLINICAL TRIAL: NCT06838351
Title: Drawing and Anxiety Study: Investigation of a Guided-Drawing and Mindfulness Intervention to Reduce Anxiety
Brief Title: Drawing and Anxiety Study
Acronym: D&A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Sarah Myruski, Assistant Research Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00021234
Record Dates: First submitted 2025-02-13; First posted 2025-02-20 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Anxiety
Keywords: anxiety; mindfulness; drawing; RSA
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Guided Drawing Group (Experimental): Participants in this group were asked to complete a guided drawing activity (~20 min). Participants were given a pencil and blank paper to use while they watched a pre-recorded video guiding them through a mindfulness and drawing activity. In the pre-recorded video, participants are instructed to draw elements of nature from exemplar photographs (e.g., leaves, twigs). The activity incorporates drawing with aspects of mindfulness meditation (i.e., being non-judgmental of thoughts and behaviors, focusing on breathing, and embodiment).
  Interventions: Behavioral: Guided Drawing Intervention
- Free Drawing Control Group (Active Comparator): In the free drawing group, participants watched a video with brief instructions and then were asked to draw whatever they would like for about 20 minutes.
  Interventions: Behavioral: Free Drawing Control
- Basic Control Group (Placebo Comparator): In the basic control group, participants were asked to complete simple paper and pencil activities (e.g., connect the dots, mazes) on their own for about 20 minutes.
  Interventions: Behavioral: Basic Control

INTERVENTIONS:
Behavioral: Guided Drawing Intervention — The guided drawing activity is a 20 minute session which integrates mindfulness and drawing elements. Participants were given a pencil and blank paper to use while they watched a pre-recorded video guiding them through a mindfulness and drawing activity. In the pre-recorded video, participants are instructed to draw elements of nature from exemplar photographs (e.g., leaves, twigs). The activity incorporates drawing with aspects of mindfulness meditation (i.e., being non-judgmental of thoughts and behaviors, focusing on breathing, and embodiment).
  Arms: Guided Drawing Group
Behavioral: Free Drawing Control — Participants are instructed to draw freely for about 20 minutes.
  Arms: Free Drawing Control Group
Behavioral: Basic Control — Participants are instructed to complete simple paper and pencil activities (e.g., mazes, connect the dots) for about 20 minutes.
  Arms: Basic Control Group

SUMMARY:
Anxiety is among the most common emotional difficulties impacting well-being, highlighting the need for approachable anxiety-reduction tools. Both mindfulness and art-based interventions have been shown to decrease anxiety symptoms. These studies integrate these approaches via a novel guided drawing intervention, and tests effects on anxiety (pre/post drawing and at one-week follow-up) and physiological regulation (respiratory sinus arrhythmia). This registration includes two separate intervention studies with similar protocols but using different samples - one consisting of adolescents ages 13 to 17.9 years, and the other consisting of adults ages 18 to 25 years. Participants complete a laboratory visit during which they complete questionnaires about their emotions and anxiety, complete pre/post measures of cardiac physiology and state anxiety, and engage in a drawing session. Participants also complete a one-week follow-up self-report of anxiety symptoms. The intervention protocol is briefly described as follows: participants in each sample are randomly assigned to one of three groups (guided drawing, free drawing control, or basic control).

DETAILED DESCRIPTION:
Materials The Screen for Adult Anxiety Related Disorders (SCAARED) is a 44-item self-report questionnaire designed for screening anxiety disorders in adulthood. Factors assessed include generalized anxiety disorder (GAD), social anxiety disorder (SAD), separation anxiety disorder, and somatic/panic/agoraphobia. Items include statements such as 'I worry about people liking me', 'People tell me that I look nervous', 'I am afraid to be alone in the house', and 'When I get anxious, I feel dizzy'. Participants indicate their response on a 3-point scale (0 = not true or hardly true ever, 1 = somewhat true or sometimes true, 2 = very true or often true). Higher scores indicate a higher likelihood of anxiety disorder(s).

State-Trait Anxiety Inventory - State Scale. The State-Trait Anxiety Inventory - State Scale (STAI-S, Spielberger et al., 1983) is a 20-item self-report questionnaire designed to assess state anxiety (current anxiety feelings). Items include statements such as 'I feel calm', 'I feel strained', and 'I am jittery'. Participants indicate their response on a 4-point scale (1 = not at all, 4 = very much so). Higher scores indicate greater state anxiety.

Participants are also asked to report on their emotion regulation difficulties as an individual difference moderator variable. The Difficulties in Emotion Regulation Scale - Short Form (DERS-SF) is an 18-item self-report questionnaire designed for assessing emotion regulation problems. Items include statements such as 'I care about what I am feeling', 'When I'm upset, I have difficulty focusing on other things', and 'When I'm upset, it takes me a long time to feel better'. Participants indicate their response on a 5-point scale (1 = almost never, 5 = almost always).

Cardiac Activity Recording and Data Processing Electrocardiogram (ECG) data was recorded using Mindware software with a sampling rate of 500 ms. Three electrodes were applied to the participants: on the distal right collarbone, the lower left rib, and the lower right rib to acquire the electrocardiogram (ECG) signal.

Experimenters manually mark the beginning and end of each episode in the cardiac data using Mindware's BioLab software. During the session, markers are placed to indicate the onset and offset of the pre-drawing period (8 minutes), the drawing session (~20 minutes; guided drawing or controls), and the post-drawing period (8 minutes). During the pre-drawing and post-drawing periods, participants complete state questionnaires (~2-3 minutes) and then remain seated until a total of 8 minutes elapsed.

Procedure

Following informed consent (~10 minutes), participants complete questionnaires to capture demographic (age, race, gender) information and individual differences in anxiety symptoms and emotion regulation difficulties (SCAARED, DERS-SF). After the questionnaires, cardiac activity monitors are applied (~15 minutes), and participants are seated to complete state questionnaires and sitting cardiac resting state (8 minutes). After completion of the pre-drawing activity portion, the experimenter returns to the observation room and prepares the drawing session to which the participant has been randomly assigned. Participants are seated in front of a desktop computer. The experimenter places two pencils, a pencil sharpener, and an 8.5" X 11" blank sketchbook on the table in front of the participant. They are read the following instructions aloud and the experimenter leaves the room:

"Next, you're going to watch a video that will walk you through a drawing exercise. You have a pencil and some paper here to use. I'll leave the room, and you will not be asked to show your drawing to anyone. The video will explain everything else you need to know. When I leave the room, press the space bar to begin the video when you are ready. I'll be back shortly after the video is done playing."

In the guided drawing video, participants are instructed to draw elements of nature from exemplar photographs (e.g., leaves, twigs). The activity incorporates drawing with aspects of mindfulness meditation (i.e., being non-judgmental of thoughts and behaviors, focusing on breathing, and embodiment). In the free drawing group, participants watch a video with brief instructions and then were asked to draw whatever they would like. In the basic control group, participants are asked to complete simple paper and pencil activities (e.g., connect the dots, mazes) on their own.

After completion of the drawing session (~20 minutes), participants again complete state questionnaires and sitting cardiac resting state (8 minutes). ECG electrodes were then removed (~5 minutes), and participants complete closing questionnaires (~10 minutes). Upon closing questionnaires, participants were given a debriefing document explaining the study's purpose and experimenters answered any questions they had (~5 minutes). Participants spend approximately 90 minutes in the laboratory.

One week after the laboratory visit, participants are sent a link, via email, to their follow-up questionnaires including SCAARED.

ELIGIBILITY:
Inclusion Criteria:

* Within the specified age range (13 to 17.9 years for adolescent version; 18 to 25 years for adult version)
* Able to speak, read and understand English

Exclusion Criteria:

* Outside the specified age range (13 to 17.9 years for adolescent version; 18 to 25 years for adult version)
* Not able to speak, read and understand English

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 275 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
State anxiety | State anxiety changes are evaluated from baseline (before drawing session) to post-drawing (i.e., about 30 minutes after baseline).
  State anxiety is measured via the State-Trait Anxiety Inventory - State Scale (STAI-S), a 20-item self-report questionnaire designed to assess state anxiety (current anxiety feelings). Participants report their state anxiety before and after the drawing session by responding to the STAI-S items (e.g., "I feel strained") using a scale from (1) not at all to (4) very much so. Sum scores are computed to quantify state anxiety before and after drawing, with possible scores ranging from 20 to 80, with higher scores indicated higher state anxiety.

SECONDARY OUTCOMES:
Anxiety Symptoms | From baseline (before drawing session) to one week later (7 days after lab visit)
  The Screen for Adult Anxiety Related Disorders (SCAARED) is a 44-item self-report questionnaire designed for screening anxiety disorders in adulthood. Items include statements such as 'I worry about people liking me', 'People tell me that I look nervous', 'I am afraid to be alone in the house', and 'When I get anxious, I feel dizzy'. Participants indicate their response on a 3-point scale (0 = not true or hardly true ever, 1 = somewhat true or sometimes true, 2 = very true or often true). Higher scores indicate a higher likelihood of anxiety disorder(s). Total anxiety symptom scores were used as a secondary outcome.

OTHER OUTCOMES:
Respiratory Sinus Arrythmia | From baseline (pre-drawing), throughout drawing session (~20 minutes), and to post-drawing (about 36 minutes after baseline start).
  Electrocardiogram (ECG) data was recorded using Mindware equipment to capture respiratory sinus arrythmia (RSA), an index of parasympathetic nervous system activity. Three electrodes were applied to the participants: on the distal right collarbone, the lower left rib, and the lower right rib to acquire the ECG signal. RSA was calculated separately for three episodes: pre-drawing, drawing, and post-drawing periods. Average RSA within each episode was used to examine within-subject change across the lab session. RSA change across episodes was computed via residual scores, with pre-drawing RSA predicting drawing RSA and post-drawing RSA. Greater residual scores reflected greater RSA augmentation, or the recruitment of parasympathetic nervous system activity during or following drawing, in comparison to baseline (pre-drawing).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Myruski, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared on the osf.oi platform. We will share scored self-report and physiological data pertinent to publications from this study.
Supporting Information: Analytic Code
Time Frame: IPD will be available upon submission of manuscripts for review and remain available via link provided by the researchers and/or corresponding author(s).
Access Criteria: Reviewers and other interested researchers will be able to access the IPD via our osf.oi repository which will be linked in any relevant publications or journal submissions.

REFERENCES:
- [Background] Kaufman, E.A., Xia, M., Fosco, G. et al. The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and Replication in Adolescent and Adult Samples. J Psychopathol Behav Assess 38, 443-455 (2016). https://doi.org/10.1007/s10862-015-9529-3
- [Background] Angulo M, Rooks BT, Gill M, Goldstein T, Sakolsky D, Goldstein B, Monk K, Hickey MB, Diler RS, Hafeman D, Merranko J, Axelson D, Birmaher B. Psychometrics of the screen for adult anxiety related disorders (SCAARED)- A new scale for the assessment of DSM-5 anxiety disorders. Psychiatry Res. 2017 Jul;253:84-90. doi: 10.1016/j.psychres.2017.02.034. Epub 2017 Feb 17. PMID 28359032
- [Background] Spielberger, C. D., Gorsuch, R. L., Lushene, R., Vagg, P. R., & Jacobs, G. A. (1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press.